CLINICAL TRIAL: NCT04172025
Title: Development of a Swiss Surveillance Database for Molecular Epidemiology of Hypervirulent and Multi-drug Resistant Pathogens
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01291; qu19Egli5
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Multiresistant Bacterial Pathogens; Virulent Bacterial Pathogens
Keywords: Epidemiology; surveillance; bacterial pathogens; Database; Genotyping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with colonization or infections with a pathogen: All patients with either colonisations or infections with either a bacterial or a viral pathogen, where whole genome sequencing data and available minimal epidemiological, demographic and clinical data
  Interventions: Diagnostic Test: Analysis of Bacterial Genome

INTERVENTIONS:
Diagnostic Test: Analysis of Bacterial Genome — genome assembly; prediction of sequence type (MLST); core genome MLST tree to rapidly compare strains within a project; core genome single nucleotide polymorphism (SNP) tree to compare all Swiss Pathogen Surveillance Platform (SPSP) strains belonging to a same species; whole genome SNP tree to compare all SPSP strains within the same species and ST;; prediction of resistance and virulence factors within pathogen submitted genomes; time trees and calculation of transmission rates, including basic reproduction number; analysis of classical epidemiological data with advanced statistical methods including machine learning.

SUMMARY:
Hypervirulent and multidrug-resistant infections are associated with significant health care costs, substantial morbidity and mortality. Therefore, the rapid recognition of outbreaks and transmissions with hypervirulent and multi-drug resistant pathogen is a key priority for infection control and public health.The main goal is to implement a shared database, connecting human and veterinary microbiology laboratories, which would allow near real-time molecular epidemiology with high spatiotemporal resolution of bacterial pathogens such as transmission and outbreak surveillance between different compartments including humans, animals and the environment in Switzerland. Investigator aims to analyze already collected encoded retrospective datasets of various pathogens by combining epidemiological data and whole genome sequences from pathogens.

DETAILED DESCRIPTION:
Hypervirulent and multidrug-resistant infections are associated with significant health care costs, substantial morbidity and mortality. Therefore, the rapid recognition of outbreaks and transmissions with hypervirulent and multi-drug resistant pathogen is a key priority for infection control and public health. For hospital epidemiologist, infectious disease and public health experts, and microbiologists the identification of an outbreak source is a first important step to establish effective counter-measurements. In Switzerland, the burden of pathogen transmission between humans, animals and the environment is substantial. The main goal is to implement a shared database, connecting human and veterinary microbiology laboratories, which would allow near real-time molecular epidemiology with high spatiotemporal resolution of bacterial pathogens such as transmission and outbreak surveillance between different compartments including humans, animals and the environment in Switzerland. Investigator aims to analyze already collected encoded retrospective datasets of various pathogens by combining epidemiological data and whole genome sequences from pathogens.

ELIGIBILITY:
Inclusion Criteria:

* All patients with either colonisations or infections with either a bacterial or a viral pathogen, where whole genome sequencing data and available minimal epidemiological, demographic and clinical data
* Pathogens included into analysis are: Multidrug-resistant bacteria include: methicillin resistant Staphylococcus aureus (MRSA), Carbapenemase- and/or extended spectrum betalactamase (ESBL)-producing Enterobacteriaceae and non-fermenting bacteria including Pseudomonas aeruginosa and Acinetobacter baumannii, Vancomycin resistant Enterococcus faecium, and others; virulent bacteria include: Neisseria meningitidis, Neisseria gonorrhoeae, Mycobacterium tuberculosis, Campylobacter spp., Salmonella spp., Legionella pneumophila, Listeria monocytogenes, and Streptococcus pneumoniae, and others; Viruses include: Influenza viruses, Measles virus, Enterovirus E68, Respiratory Syncytial Virus and others.

Exclusion Criteria:

* Decline to sign a general consent or any other declining statement against using data for research purposes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: • All patients with either colonisations or infections with either a bacterial or a viral pathogens including the below listed pathogens from participating centers in Switzerland.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of transmission clusters based on genetic similarity. | Onetime identification at baseline
  Identification of transmission clusters based on genetic similarity. With focus on whole genome sequencing.

SECONDARY OUTCOMES:
Detection of Genotypic Resistance | Onetime identification at baseline
  Detection of Genotypic Resistance (in-vitro antibiotic susceptibility test (AST) based on measuring minimum inhibitory concentration (MIC) or zone diameter (ZD))

CONTACTS AND LOCATIONS:
Overall Officials: Hans Hirsch, Prof. Dr., Principal Investigator — Biozentrum, University of Basel
Locations (5):
- Switzerland (5):
  - University Hospital Basel, Basel
  - University of Bern, Bern
  - University Hospital Geneva, Geneva
  - University Hospital Lausanne CHUV, Lausanne
  - University of Zurich, Zurich

REFERENCES:
- [Background] Cassini A, Hogberg LD, Plachouras D, Quattrocchi A, Hoxha A, Simonsen GS, Colomb-Cotinat M, Kretzschmar ME, Devleesschauwer B, Cecchini M, Ouakrim DA, Oliveira TC, Struelens MJ, Suetens C, Monnet DL; Burden of AMR Collaborative Group. Attributable deaths and disability-adjusted life-years caused by infections with antibiotic-resistant bacteria in the EU and the European Economic Area in 2015: a population-level modelling analysis. Lancet Infect Dis. 2019 Jan;19(1):56-66. doi: 10.1016/S1473-3099(18)30605-4. Epub 2018 Nov 5. PMID 30409683
- [Background] Daxboeck F, Budic T, Assadian O, Reich M, Koller W. Economic burden associated with multi-resistant Gram-negative organisms compared with that for methicillin-resistant Staphylococcus aureus in a university teaching hospital. J Hosp Infect. 2006 Feb;62(2):214-8. doi: 10.1016/j.jhin.2005.07.009. Epub 2005 Oct 27. PMID 16257092
- [Background] Egli A, Blanc DS, Greub G, Keller PM, Lazarevic V, Lebrand A, Leib S, Neher RA, Perreten V, Ramette A, Schrenzel J, Stephan R, Wagner K, Wuethrich D, Xenarios I. Improving the quality and workflow of bacterial genome sequencing and analysis: paving the way for a Switzerland-wide molecular epidemiological surveillance platform. Swiss Med Wkly. 2018 Dec 15;148:w14693. doi: 10.4414/smw.2018.14693. eCollection 2018 Dec 3. PMID 30552858
- [Background] Ford L, Carter GP, Wang Q, Seemann T, Sintchenko V, Glass K, Williamson DA, Howard P, Valcanis M, Castillo CFS, Sait M, Howden BP, Kirk MD. Incorporating Whole-Genome Sequencing into Public Health Surveillance: Lessons from Prospective Sequencing of Salmonella Typhimurium in Australia. Foodborne Pathog Dis. 2018 Mar;15(3):161-167. doi: 10.1089/fpd.2017.2352. Epub 2018 Jan 16. PMID 29336594
- [Background] Meinel DM, Kuehl R, Zbinden R, Boskova V, Garzoni C, Fadini D, Dolina M, Blumel B, Weibel T, Tschudin-Sutter S, Widmer AF, Bielicki JA, Dierig A, Heininger U, Konrad R, Berger A, Hinic V, Goldenberger D, Blaich A, Stadler T, Battegay M, Sing A, Egli A. Outbreak investigation for toxigenic Corynebacterium diphtheriae wound infections in refugees from Northeast Africa and Syria in Switzerland and Germany by whole genome sequencing. Clin Microbiol Infect. 2016 Dec;22(12):1003.e1-1003.e8. doi: 10.1016/j.cmi.2016.08.010. Epub 2016 Aug 30. PMID 27585943
- [Background] Phodha T, Riewpaiboon A, Malathum K, Coyte PC. Excess annual economic burdens from nosocomial infections caused by multi-drug resistant bacteria in Thailand. Expert Rev Pharmacoecon Outcomes Res. 2019 Jun;19(3):305-312. doi: 10.1080/14737167.2019.1537123. Epub 2018 Oct 19. PMID 30321493
- [Background] Seth-Smith HMB, Casanova C, Sommerstein R, Meinel DM, Abdelbary MMH, Blanc DS, Droz S, Fuhrer U, Lienhard R, Lang C, Dubuis O, Schlegel M, Widmer A, Keller PM, Marschall J, Egli A. Phenotypic and Genomic Analyses of Burkholderia stabilis Clinical Contamination, Switzerland. Emerg Infect Dis. 2019 Jun;25(6):1084-1092. doi: 10.3201/eid2506.172119. PMID 31107229
- [Background] Sommerstein R, Fuhrer U, Lo Priore E, Casanova C, Meinel DM, Seth-Smith HM, Kronenberg A; Anresis; Koch D, Senn L, Widmer AF, Egli A, Marschall J; Swissnoso. Burkholderia stabilis outbreak associated with contaminated commercially-available washing gloves, Switzerland, May 2015 to August 2016. Euro Surveill. 2017 Dec;22(49):17-00213. doi: 10.2807/1560-7917.ES.2017.22.49.17-00213. PMID 29233255
- [Background] Stucki D, Ballif M, Egger M, Furrer H, Altpeter E, Battegay M, Droz S, Bruderer T, Coscolla M, Borrell S, Zurcher K, Janssens JP, Calmy A, Mazza Stalder J, Jaton K, Rieder HL, Pfyffer GE, Siegrist HH, Hoffmann M, Fehr J, Dolina M, Frei R, Schrenzel J, Bottger EC, Gagneux S, Fenner L. Standard Genotyping Overestimates Transmission of Mycobacterium tuberculosis among Immigrants in a Low-Incidence Country. J Clin Microbiol. 2016 Jul;54(7):1862-1870. doi: 10.1128/JCM.00126-16. Epub 2016 May 18. PMID 27194683
- [Background] Walker TM, Merker M, Knoblauch AM, Helbling P, Schoch OD, van der Werf MJ, Kranzer K, Fiebig L, Kroger S, Haas W, Hoffmann H, Indra A, Egli A, Cirillo DM, Robert J, Rogers TR, Groenheit R, Mengshoel AT, Mathys V, Haanpera M, Soolingen DV, Niemann S, Bottger EC, Keller PM; MDR-TB Cluster Consortium. A cluster of multidrug-resistant Mycobacterium tuberculosis among patients arriving in Europe from the Horn of Africa: a molecular epidemiological study. Lancet Infect Dis. 2018 Apr;18(4):431-440. doi: 10.1016/S1473-3099(18)30004-5. Epub 2018 Jan 8. PMID 29326013
- [Background] Ward DV, Hoss AG, Kolde R, van Aggelen HC, Loving J, Smith SA, Mack DA, Kathirvel R, Halperin JA, Buell DJ, Wong BE, Ashworth JL, Fortunato-Habib MM, Xu L, Barton BA, Lazar P, Carmona JJ, Mathew J, Salgo IS, Gross BD, Ellison RT. Integration of genomic and clinical data augments surveillance of healthcare-acquired infections. Infect Control Hosp Epidemiol. 2019 Jun;40(6):649-655. doi: 10.1017/ice.2019.75. Epub 2019 Apr 23. PMID 31012399
- [Background] Wassilew N, Seth-Smith HM, Rolli E, Fietze Y, Casanova C, Fuhrer U, Egli A, Marschall J, Buetti N. Outbreak of vancomycin-resistant Enterococcus faecium clone ST796, Switzerland, December 2017 to April 2018. Euro Surveill. 2018 Jul;23(29):1800351. doi: 10.2807/1560-7917.ES.2018.23.29.1800351. PMID 30043725
- [Background] Wuthrich D, Gautsch S, Spieler-Denz R, Dubuis O, Gaia V, Moran-Gilad J, Hinic V, Seth-Smith HM, Nickel CH, Tschudin-Sutter S, Bassetti S, Haenggi M, Brodmann P, Fuchs S, Egli A. Air-conditioner cooling towers as complex reservoirs and continuous source of Legionella pneumophila infection evidenced by a genomic analysis study in 2017, Switzerland. Euro Surveill. 2019 Jan;24(4):1800192. doi: 10.2807/1560-7917.ES.2019.24.4.1800192. PMID 30696527